CLINICAL TRIAL: NCT00381511
Title: Objective Assessment of Pulmonary Embolism Can be Deferred Without Increased Risk
Brief Title: Deferment of Imaging for Pulmonary Embolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3090A-101657
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-09

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism,; deferred diagnosis,; protective anticoagulation; anticoagulants
MeSH Terms: conditions — Pulmonary Embolism | interventions — Heparin, Low-Molecular-Weight

INTERVENTIONS:
Drug: low molecular weight heparin

SUMMARY:
Background. Management of patients with suspected Pulmonary Embolism (PE) is problematic if diagnostic imaging is not available. Pretest Clinical Probability (PCP) and D-dimer (D-d) assessment were shown to be useful to identify those high risk patients for whom empirical, protective anticoagulation is indicated.

To evaluate whether PCP and D-d assessment, together with the use of low molecular weight heparins (LMWHs), allow objective appraisal of PE to be deferred for up to 72 hours, we planned to prospectively evaluate consecutive patients with suspected PE.

Methods. In case of deferment of diagnostic imaging for PE, patients identified at high-risk (those with high PCP or moderate PCP and positive D-d), receive a protective full-dose treatment of LMWH; the remaining patients will be discharged without anticoagulant. All patients will be scheduled to undergo objective tests for PE within 72 hours. Standard antithrombotic therapy will be then administered when diagnostic tests confirmed Venous ThromboEmbolism (VTE).

DETAILED DESCRIPTION:
Introduction Pulmonary Embolism (PE), the most serious complication of Deep Vein Thrombosis (DVT), is a relatively common and potentially fatal disease. Its diagnosis usually requires multiple approaches based on diagnostic imaging such as ventilation/perfusion lung scanning (V/Q) or Computed Tomography (CT). However, the performance of such imaging cannot immediately be performed in case of night or week-end referral; in this situation, attending physicians have to decide whether to treat incompletely assessed patients or to hospitalise them until confirmatory tests can be carried out. In lack of guidelines, empirical protective anticoagulation with Low Molecular Weight Heparins (LMWH), drugs showing a more favourable pharmacodynamic profile in comparison to UnFractionated Heparins (UFH), is usually given to patients. However, no clear-cut information is available about the need of such anticoagulation, its dosage and duration, or the time over which deferral of diagnostic procedures can be considered as safe. It seems more appropriate and safer, though, a management based on a preliminary evaluation of the actual risk of thrombosis.

We have recently demonstrated that in patients clinically suspected of venous thromboembolism, Pre-test Clinical Probability (PCP), D-dimer and the use of LMWH can be safely used for delaying diagnostic tests for up 72 hours (Siragusa S et al. Arch Intern Med 2004;164:2477). Our paper was mainly focused to patients suspected of Deep Vein Thrombosis (about 80% of the patients' cohort) which are considered a category at lower risk for complications than PE patients.

Critically, data are lacking to guide the management of patients clinically suspected of having PE who cannot undergo immediate diagnostic imaging.

We plan to perform a prospective clinical trial aimed at evaluating whether data derived from PCP and D-dimer testing, together with the use of LMWHs, permit safe management of patients with suspected PE when objective assessment is not available.

Materials and Methods Patient Population Out-patients presenting with suspected acute PE, when diagnostic imaging were not immediately available (during nights or week-ends), will be considered eligible for the study. The study will be conducted in three Institutions (University Hospital AOUP "Paolo Giaccone" of Palermo, IRCCS Policlinico S. Matteo, Italy and IRCCS Ospedale Maggiore di Milano, Italy) with the same protocol. Exclusion criteria included the following: 1) life-threatening conditions, or serious co-morbidities that required immediate hospitalisation ; 2) relapse of a previously documented PE episode; 3) current use of oral anticoagulant therapy; 4) history of bleeding or any other contraindication to heparin; 5) age younger than 18 years; 6) life expectancy of less than 3 months; 7) refusal to give informed consent.

Algorithm of intervention Patients will be evaluated and managed according to the clinical assessment protocol. PCP for PE will be assessed first (using a previously reported clinical model, followed by the D-dimer test.

Patients considered at "low-risk", in case of low PCP or moderate PCP with a negative D-dimer test result, will be discharged without anticoagulant therapy. Conversely, patients with moderate PCP and a positive D-dimer test or with high PCP , will be considered as being at "high risk" and will receive therapeutic doses of LMWHs as 'protective anticoagulation'. Physicians have indeed the option of admitting patients to the hospital irrespective of PCP and D-dimer test results. All patients, either managed as in or out-patients, havo to undergo diagnostic imaging within 72 hours of PCP and D-dimer test assessment.

Diagnostic assessment protocol for PE Diagnosis of PE will be assessed as described; briefly, all patients will undergo Ventilation-perfusion (V/Q) lung scanning or lung CT within 72 hours from the patient referral. In case of not diagnostic imaging, patients undergo ultrasonography of the lower limbs. Patients weill be diagnosed as having PE if they have a high-probability V/Q scan or an abnormal imaging result showing venous thrombi. All diagnostic tests will be performed by operators unaware of D-d assay results or PCP assessment. In cases of a positive diagnostic imaging test results, patients will be managed accordingly and they will receive full dose of anticoagulants.

Blood drawn for the D-dimer assay will be mixed with tri-sodium citrate (1 vol) and tested by technicians unaware of other test results. We will use a semi-quantitative latex assay (Dimertest®, Dade Behring, Deerfield Ill) performed as described.

Follow-Up Patients will be monitored for 2 periods of follow-up: short-term and long-term. Short-term follow-up is defined as the time between patient referral and the completion of the diagnostic procedures (within 72 hours). Patients will be trained to return or to contact physicians during this period in case of: 1) worsening of respiratory symptoms; 2) signs and symptoms suggestive of developing deep venous thrombosis of the legs; 3) major and minor bleeding during protective anticoagulation; 4) any other reason for hospitalisation due to VTE-related symptoms.

Long-term follow-up (3 months) is used to record the incidence of PE in those patients for whom this diagnosis will be ruled out.

At any follow up time, in case of signs or symptoms suggestive of the aforementioned events, patients will undergo objective assessment through imaging.

Statistic analysis We estimate that the primary event rate (PE and major bleeding) during the short-term follow-up would be less than 2%. We plan to include a sufficient number of patients to ensure that the upper limits of the 95% Confidence Intervals (CI) were less than 2.5%. This resulted in a projected sample size of at least 300 patients.

The rate of occurrence of any thromboembolic event during the short- or long-term follow-up will be determined and 95% CI will be calculated. The proportion of patients who developed VTE in each PCP group and the relative 95% CI will be determined, as were the proportions of patients who develope events during the long-term follow up. Paired "t" and Pearson 2 tests were used as indicated; P < .05% (2-tailed) was considered statistically significant. Diagnostic accuracy of D-dimer assessment will be calculated in terms of sensitivity, specificity, and positive and negative predictive values with corresponding 95% CIs (9).

ELIGIBILITY:
Inclusion Criteria:

* Out-patients presenting with suspected acute PE, when diagnostic imaging are not immediately available (during nights or week-ends), are considered eligible for the study.

Exclusion Criteria:

* life-threatening conditions, or serious co-morbidities that required immediate hospitalisation ;
* relapse of a previously documented PE episode;
* current use of oral anticoagulant therapy;
* history of bleeding or any other contraindication to heparin;
* age younger than 18 years;
* life expectancy of less than 3 months;
* refusal to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1999-01; Study Completion 2004-04

PRIMARY OUTCOMES:
Recurrent venous thromboembolism
major bleeding
death

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Siragusa, MD, Principal Investigator — University Hospital of Palermo